CLINICAL TRIAL: NCT06201442
Title: Profiling of Abnormal Knee Joint Loading to Reduce Risk of Post-Traumatic Knee Osteoarthritis Following Anterior Cruciate Ligament Reconstruction
Brief Title: Post-Traumatic Knee Osteoarthritis Following Anterior Cruciate Ligament Reconstruction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S65257
Record Dates: First submitted 2023-01-26; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-08

CONDITIONS: Anterior Cruciate Ligament Injuries; Post-Traumatic Osteoarthritis of Knee
Keywords: ACLR; Anterior cruciate ligament injury; PTOA; post-traumatic knee osteoarthritis; KJPM; knee joint pathomechanics
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients undergoing unilateral Anterior Cruciate Ligament Reconstruction (ACLR): 4 - 5 visits: Clinical examination, magnetic resonance imaging (MRI), 3D motion analysis, Strength assessment, EOS radiography (full leg X-ray scan), X-ray scan knee, Blood sample, Questionnaires and Activity monitoring.
  Interventions: Other: Imaging - magnetic resonance imaging (MRI); Other: Blood sampling; Other: Assessment of functionality and strength; Other: Activity monitoring; Other: Imaging - x-ray scan (RX); Behavioral: Questionnaires
- Healthy controls without previous Anterior Cruciate Ligament (ACL) injury: 2 visits: Clinical examination, MRI, 3D motion analysis, Strength assessment, EOS radiography, X-ray scan knee, Blood sample, Questionnaires and Activity monitoring.
  Interventions: Other: Imaging - magnetic resonance imaging (MRI); Other: Blood sampling; Other: Assessment of functionality and strength; Other: Activity monitoring; Other: Imaging - x-ray scan (RX); Behavioral: Questionnaires

INTERVENTIONS:
Other: Imaging - magnetic resonance imaging (MRI) — MRI knee - not standard of care
Other: Blood sampling — blood sample taken and analysis - not standard of care
Other: Assessment of functionality and strength — Movements and posture Analysis Laboratory Leuven measurement (3D motion analysis) and Biodex measurement - not standard of care
Other: Activity monitoring — Actigraph measurement- not standard of care
Other: Imaging - x-ray scan (RX) — RX Knee and EOS radiography full leg - not standard of care
Behavioral: Questionnaires — Patient reported outcomes (PROMS)

SUMMARY:
The purpose of this trial is to define knee joint pathomechanics (KJPM) in the first 2 years after ACL reconstruction (ACLR) and relate these KJPM with changes in articular cartilage morphology and quality.

DETAILED DESCRIPTION:
This research project is a longitudinal prospective study. The investigators aim to define the KJPM longitudinally in the first 2 years following ACLR. The investigators relate these KJPM, combined with the cumulative mechanical exposure, to changes in articular cartilage/joint surface morphology and quality. To investigate the loading pattern on the knee joint, daily activities like walking, running and climbing stairs will be performed by the participants.

The overall goal of this research project is to investigate whether KJPM are related with early cartilage degeneration. This is a first major step towards reducing the risk for post-ACLR onset of Post-Traumatic Knee Osteoarthritis (PTOA).

Two work packages (WP) can be separated, that each have a separate aim:

WP1: The first aim of this WP (WP1.A) is to profile longitudinal changes in knee contact forces (KCFs) and knee contact pressure (KCP) distribution of the articular cartilage in the first 2 years following ACLR. Second, in WP1.B, the investigators will identify multivariate proxies of KCFs (and KCP) to improve clinical translation (for example by facilitating the development of prognostic tools for verifying KJPM in real life).

WP2: the second aim is to establish the relationship between KJPM at different time points following ACLR and (changes in) articular cartilage morphology and quality (WP2.A). Furthermore, the investigators will compare the biomechanical profile of "fast PTOA progressors" with "fast non-traumatic early osteoarthritis progressors" (WP2.B).

ELIGIBILITY:
Inclusion Criteria (healthy volunteers):

* Age: 18-35 years
* No previous anterior cruciate ligament (ACL) injury
* Body Mass Index (BMI) between 18-30
* Regular physical activity (active during work or practicing sports regularly)
* Signed informed consent to participate

Exclusion Criteria (healthy volunteers):

* Major injuries to the lower extremities with absence from sports or daily life activities longer than 2 weeks or that required surgery, less than 6 months before participation
* Pre-existing arthritic disease including inflammatory or infectious arthritis

Inclusion Criteria (ACL patients):

* Age: 18-35 years
* ACL tear which is recently reconstructed or will be reconstructed after enrollment in the current study (the reconstruction will take place within 6 months after injury) with a Hamstring autograft
* BMI between 18-30
* Regular physical activity (active during work or practicing sports regularly)
* Signed informed consent to participate

Exclusion Criteria (ACL patients):

* Major injuries to the lower extremities with absence from sports or daily life activities longer than 2 weeks or that required surgery, less than 6 months before participation
* Pre-existing arthritic disease including inflammatory or infectious arthritis
* Image based confirmation of local cartilage lesion grade 4 or major cartilage damage (Kellgren & Lawrence > 2)
* Medial collateral ligament damage (> grade 2)
* Intra-articular knee fractures
* Menisectomy with <80% remnant

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adult patients up until 35 years old with an ACL reconstruction (recruited at the outpatient clinic) Healthy controls (community sample recruited)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-11-23 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Knee contact forces (KCF) will be measured using a 3D motion analysis system | 2 years
  The goal is to profile longitudinal changes in KCFs of the articular cartilage.
  Using a 3D motion analysis system (Vicon, Oxford Metrics, UK), marker trajectories, ground reaction forces (AMTI, MA, USA) and muscle activations (Wireless EMG Cometa, Italy) will be measured. Subsequently a musculoskeletal modelling workflow in OpenSim will be used to calculate Knee contact forces (KCF) of the articular cartilage.
Knee contact pressures (KCP) will be measured using a 3D motion analysis system | 2 years
  Using a 3D motion analysis system (Vicon, Oxford Metrics, UK), marker trajectories, ground reaction forces (AMTI, MA, USA) and muscle activations (Wireless EMG Cometa, Italy) will be measured. Subsequently a musculoskeletal modelling workflow in OpenSim will be used to calculate Knee contact pressures (KCP) of the articular cartilage.
The patient-specific cartilage thickness distribution. | 2 years
  The cartilage thickness will be measured using the semi-automatic segmentation from the high-resolution images (3D-FSE) of the tibiofemoral cartilage.
The patient-specific tibiofemoral cartilage quality. | 2 years
  The cartilage quality will be examined using compositional measures such as T1rho, T1p and T2 relaxation time.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Verschueren, PhD, Principal Investigator — KU Leuven
Locations (1):
- Faculty of Kinesiology and Rehabilitation Sciences, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The full pseudonymized dataset will be made available in RDR (KU Leuven tool) and will be shared upon written request after approval of the PI, for clearly defined research purposes.
  Pseudonymized data and documentation will be available on request in RDR.
  Data sharing can only happen when it is not for commercial use or it doesn't reveal the identity of the participants. Data will always be pseudonimized.
Supporting Information: Study Protocol, CSR
Time Frame: Upon publication of the research results and for an undetermined period of time.
Access Criteria: Data sharing can only happen when it is not for commercial use or it doesn't reveal the identity of the participants. Data will always be pseudonimized. A written request has to be submitted to the PI.